CLINICAL TRIAL: NCT01043965
Title: Evaluation of Myocardial Perfusion and Microvascular Reserve in Real-time Utilizing Myocardial Contrast Echocardiography in Type 2 Diabetes.
Brief Title: Myocardial Perfusion in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Wilson Mathias Jr, Heart Institute - Sao Paulo - Brazil
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0925; nata925 (Other Grant/Funding Number: 05/57793-6R)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2005-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Myocardial perfusion imaging; Heart diseases; Echocardiography; Endothelium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Heart Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes (Active Comparator): Type 2 diabetes patients without obstructive coronary disease. Interventional group: lifestyle changes and treatment with metformin.
  Interventions: Drug: Metformin
- Control (No Intervention): Control group - normal, healthy individuals.

INTERVENTIONS:
Drug: Metformin — Metformin 850mg
  Other Names: Glucophage
  Arms: Diabetes

SUMMARY:
The investigators aimed to evaluate microvascular circulation with novel method: real-time myocardial contrast echocardiography in patients with type 2 diabetes and normal coronary arteries.

Myocardial blood flow reserve will be determined by quantitative contrast Stress echocardiography. Diabetic individuals will be evaluate in a decompensated state (Phase 1) and after optimization of medical treatment four months later (Phase 2).

DETAILED DESCRIPTION:
Early stages of epicardial atherosclerosis in patients with type 2 diabetes are associated with an impairment in endothelium-dependent dilation of the coronary microvasculature, indicating that the pathophysiological consequences of atherosclerosis may extend into the coronary microcirculation.

The investigators will evaluate three parameters of myocardial quantification with contrast Stress echocardiography and correlate with HbA1C levels.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Normal echocardiogram
* Absence of obstructive epicardial coronary disease

Exclusion Criteria:

* Obstructive coronary disease
* Heart valve disease
* COPD
* Cardiac Arrhythmias
* Cardiomyopathy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
myocardial blood flow velocity, myocardial blood flow reserve | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Mathias Jr, Md, PhD, Study Director — Heart Institute - Sao Paulo - Brazil